CLINICAL TRIAL: NCT01687634
Title: Home Visiting for Low Income, Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: W.K. Kellogg Foundation (Other); Center for HIV Identification, Prevention, and Treatment Services (Unknown)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Director, Global Center for Children and Families, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P3018725
Record Dates: First submitted 2012-09-07; First posted 2012-09-19 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pregnant Women; Nutrition During Pregnancy; Breast Feeding; Newborns
Keywords: pregnancy; home healthcare visits; breast feeding; nutrition; community health workers
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-home Mentor Mother visits (Experimental): Pregnant women will receive twice-monthly in-home (or telephone) visits from a Mentor Mother who will provide information about pregnancy, breastfeeding, nutrition, and infant care.
  Interventions: Behavioral: In-home Mentor Mother visits
- Health Information Mailings (Experimental): Pregnant women will receive twice-monthly mailings that will provide information about pregnancy, breastfeeding, nutrition, and infant care.
  Interventions: Behavioral: Health Information Mailings

INTERVENTIONS:
Behavioral: In-home Mentor Mother visits — Pregnant women will receive twice-monthly in-home (or telephone) visits from a Mentor Mother who will provide information about pregnancy, breastfeeding, nutrition, and infant care.
  Arms: In-home Mentor Mother visits
Behavioral: Health Information Mailings — Pregnant women will receive twice-monthly mailings that will provide information about pregnancy, breastfeeding, nutrition, and infant care.
  Arms: Health Information Mailings

SUMMARY:
In the Pico-Union/Koreatown community of Los Angeles investigators are designing a preventive health care model that increases the opportunities for families to make healthy choices -- in their homes, schools & communities. The project's key element is: Lay community health workers (paraprofessionals) - Mentor Mothers (MM) (promotoras) - who make home visits to pregnant mothers & newly-delivered mothers who have agreed to participate in the research study.

Investigators hope to achieve the following outcomes: 1) lower maternal BMI at 6 months post-birth; 2) longer duration of breastfeeding; 3) less alcohol, smoking, and drug use during pregnancy; and 4) increased and consistent prenatal and postnatal healthcare adherence.

Investigators will implement the study with 6 MMs, who will maintain an average caseload of 16 women each across an 18-month period. Each participant will be visited (or receive the intervention by telephone) twice per month.

Separate Assessment Team members will conduct assessments at: Baseline, within a week of birth of the target child, and 6 months from birth.

DETAILED DESCRIPTION:
After participant mothers have been recruited, screened, and consented into the study, each woman will be contacted by a member of the Assessment Team to schedule the in-home Baseline Assessment. The Baseline Assessment will take approximately 90 minutes to complete.

Follow-up Assessments will take place: within a week of delivery and 6 months after delivery. Interviews will be audio-recorded for quality assurance purposes. The domains of the Follow-up Assessments will be 1) maternal weight, height, and eating and exercise routines; 2) feeding routines, style, and frequency; 3) substance use; and 4) adherence to health care prenatally and postnatally, immunizations, and illnesses for mothers and babies. Secondarily, investigators will assess the mother's pregnancy, general health, mental health, social support, the father of the child, use of alternative medicine and health care, reproductive health, HIV, relationships and violence, baseline knowledge of antenatal health, baseline knowledge of delivery health, and baseline stated future plans.

All in-home interviews will take place in a private room or area of the participant's home. If an in-home interview is not practical or appropriate for any reason, the interviewer will conduct the interview at the Robert F. Kennedy Community Schools campus, UCLA, or another site.

Assessment team in-home interviews will be audio-recorded for quality assurance & supervision purposes. Telephone interviews will not be audio-recorded.

----------------------------------------------------

IN-HOME (OR TELEPHONE) MENTOR MOTHER INTERVENTION VISITS:

Each participant will be assigned to a Mentor Mother (MM). Participants will receive a series of twice-monthly, pre- and post-natal, in-home (or telephone call) intervention visits, for the study period of 12 months, from her assigned MM. The MM will measure the mother's height & weight at each intervention home visit, then proceed to deliver one of the Intervention Topics (e.g. nutrition, substance use awareness, infant development etc.). After the baby is born, the Mentor Mother will continue to record the mother's weight and height, and will also measure and weigh the infant, entering that data into the study mobile phone. These intervention visits (or phone calls) will last for approximately 1 hour each. The MM will address any concerns or questions the mother has, provide referrals to community resources as necessary, and leave handouts for the participant mother based on the day's intervention topic and/or the participant mother's questions that day.

----------------------------------------------------

HEALTH INFORMATION MAILINGS:

Pregnant women will receive twice-monthly mailing that will provide information about pregnancy, breastfeeding, nutrition, and infant care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Currently pregnant;
* Living in the Pico/Union Koreatown community;
* Ability to provide informed consent;
* Speaks English or Spanish

Exclusion Criteria:

* Under 18 years of age;
* Not currently pregnant;
* Not living in the Pico/Union Koreatown community;
* Unable to provide informed consent;
* Does not speak English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2012-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | Six months post-birth
Maternal BMI | Six months post-birth

SECONDARY OUTCOMES:
Alcohol, tobacco, and drug use in pregnancy | one week post-birth
World Health Organization infant age-standardized weight, length, weight-for-length, and head circumference | one week post-birth
World Health Organization infant age-standardized weight, length, weight-for-length, and head circumference | six months post-birth
Adherence to prenatal clinic visits | one week post-birth
Adherence to well-baby clinic visits | six months post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram-Borus, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Robert F. Kennedy Schools, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be be made available on the Center for HIV Identification, Prevention, and Treatment Services (CHIPTS) website.

REFERENCES:
- [Derived] Rotheram-Fuller EJ, Swendeman D, Becker KD, Daleiden E, Chorpita B, Harris DM, Mercer NT, Rotheram-Borus MJ. Replicating Evidence-Based Practices with Flexibility for Perinatal Home Visiting by Paraprofessionals. Matern Child Health J. 2017 Dec;21(12):2209-2218. doi: 10.1007/s10995-017-2342-8. PMID 28755042
- [Derived] Rotheram-Fuller E, Swendeman D, Becker K, Daleiden E, Chorpita B, Youssef MK, Rotheram-Borus MJ. Adapting Current Strategies to Implement Evidence-Based Prevention Programs for Paraprofessional Home Visiting. Prev Sci. 2017 Jul;18(5):590-599. doi: 10.1007/s11121-017-0787-z. PMID 28451922